CLINICAL TRIAL: NCT03721068
Title: A Phase I Study of Autologous Activated T-Cells Expressing a 2nd Generation GD2 Chimeric Antigen Receptor, IL-15, and iCaspase9 Safety Switch Administered To Patients With Relapsed/Refractory Neuroblastoma or Relapsed/Refractory Osteosarcoma
Brief Title: Study of CAR T-Cells Targeting the GD2 With IL-15+iCaspase9 for Relapsed/Refractory Neuroblastoma or Relapsed/Refractory Osteosarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Bellicum Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1743-ATL; K12CA120780 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma; Osteosarcoma
Keywords: Autologous Chimeric Antigen Receptor (CAR) T Cells; Interleukin (IL)-15; Disialoganglioside (GD2); Caspase 9; Pediatric; Rimiducid; AP1903; modified T cells; CAR T
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma; Gaucher Disease | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iC9.GD2.CAR.IL-15 T-cells (Experimental): The continuous reassessment method (CRM) will be used to estimate the maximum-tolerated dose (MTD) of cells that to be given in dose escalation cohorts comprised of 2-6 subjects. The final MTD will be the dose with estimated probability of dose limiting toxicity (DLT) closest to the target toxicity rate of 20%. Three cell doses will be evaluated: 0.5 x 10^6 cells/kg, 1.0 x 10^6 cells/kg, 1.5 x 10^6 cells/kg. Cohort enrollment will be staggered and each subject must complete at least 2 weeks of the cell treatment without incident of DLT before another subject can be enrolled at that dose level. A minimum of two subjects must complete the 4-week post-infusion DLT period before enrollment at the next higher dose level will be considered. If dose level 1 is determined to be above a tolerable dose, de-escalation would occur to dose level -1 where subjects would receive 0.25 x 10^6 cells/kg.
  Interventions: Biological: iC9.GD2.CAR.IL-15 T-cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: iC9.GD2.CAR.IL-15 T-cells — Three dose levels are being evaluated: 0.5 x 10^6, 1.0 x 10^6, 1.5 x 10^6
Drug: Cyclophosphamide — 500 mg/m^2 IV dose on days 1-2 for lymphodepletion prior to cell infusion
Drug: Fludarabine — 30 mg/m^2 IV dose on days 1-4 for lymphodepletion prior to cell infusion

SUMMARY:
The body has different ways of fighting infections and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are molecules that fight infections and protect your body from diseases caused by bacteria and toxic substances. Antibodies work by sticking to those bacteria or substances, which stops them from growing and causing bad effects. T cells are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected. Both antibodies and T cells have been used to treat patients with cancers. They both have shown promise, but neither alone has been enough to cure most patients.

This multicenter study is designed to combine both T cells and antibodies in order to create a more effective treatment. The treatment that is being researched is called autologous T lymphocyte chimeric antigen receptor cells (CAR) cells targeted against the disialoganglioside (GD2) antigen that express Interleukin (IL)-15, and the inducible caspase 9 safety switch (iC9), also known as iC9.GD2.CAR.IL-15 T cells.

DETAILED DESCRIPTION:
In previous studies, it has been shown that when T cells have part of an antibody attached to them, they are better at recognizing and killing cancer cells. The antibody that will be used in this study is called anti-GD2. This antibody floats around in the blood and can detect and stick to cancer cells called neuroblastoma cells because they have a substance on the outside of the cells called GD2. For this study, the anti-GD2 antibody has been changed so that instead of floating freely in the blood, it is now joined to the T cells. However, it is unknown how long the iC9.GD2.CAR.IL-15 T cells last in the body, so their chances of fighting cancer cells are not well known.

To improve the tumor-fighting power of GD2-CAR-T cells, two additional components were added to these cells. The IL-15 gene was added so that the GD2-CAR-T cells can attack tumor cells more effectively. Interleukin-15 (IL-15) is a chemical that cells use to communicate with one another. Other research using IL-15 in combination with CAR-T cells has shown there is an increase in the body's ability to allow the CAR-T cells to survive and grow in the body. The iC9 gene was added as an "off switch" so it can stop the activity of the GD2-CAR-T cells if there are any serious bad side effects. Bad side effects seen previously in patients receiving the GD2 antibody alone include pain. In this study, the "stop switch" can be used to turn off the GD2-CAR-T cells if you experience intense pain that does not respond to normal pain treatments.

The study will enroll a minimum of 10 adult subjects and 10 pediatric subjects; all subjects will undergo lymphodepletion chemotherapy prior to the cell infusion as outlined in the protocol.

ELIGIBILITY:
All clinical and laboratory data required for determining eligibility must be available in the subject's medical/research record which will serve as the source document.

Because of the nature of iC9.GD2.CAR.IL-15 T cell product preparation, subjects will be assessed for initial study enrollment eligibility (prior to cell procurement) and then will have to meet criteria prior to starting lymphodepletion and prior to T cell infusion.

Inclusion Criteria for the Study:

1. Written HIPAA authorization signed by legal guardian.
2. Adequate performance status as defined by Lansky or Karnofsky performance status of ≥ 60 (Lansky for <16 years of age).
3. Life expectancy ≥12 weeks.
4. Histological confirmation of neuroblastoma or ganglioneuroblastoma at initial diagnosis. Bone marrow samples are acceptable as confirmation of neuroblastoma, confirmation of osteosarcoma at diagnosis
5. High-risk neuroblastoma with persistent/refractory or relapsed disease, defined as:

   1. First or greater relapse of neuroblastoma following completion of aggressive multi-drug frontline therapy.
   2. First episode of progressive neuroblastoma during aggressive multi-drug frontline therapy. Persistent/refractory neuroblastoma as defined by less than a complete response by the revised International Neuroblastoma Response Criteria (INRC) at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocol (such as A3973 or ANBL0532).
   3. Patients must be diagnosed with high risk neuroblastoma at initial diagnosis or if non-high risk at time of initial diagnosis must have had evidence of metastatic progression when >18 months of age as defined in the protocol or relapsed or refractory osteosarcoma that is not responsive to standard treatment.
6. Measurable or evaluable disease per Revised INRC for subjects with neuroblastoma or measurable disease by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 criteria for subjects with osteosarcoma.
7. Adequate central nervous system function as defined by:

   1. No known Central Nervous System ( CNS) disease
   2. No seizure disorder requiring antiepileptic drug therapy

Exclusion Criteria for the Study Subjects meeting any of the following exclusion criteria will not be able to participate in this study (procurement, lymphodepletion, and cell infusion).

1. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
2. Has a known additional malignancy that is active and/or progressive requiring treatment.
3. History of hypersensitivity reactions to murine protein-containing products.
4. History of hypersensitivity to cyclophosphamide or fludarabine.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2030-05-19 (Estimated); Study Completion 2044-06-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of iC9.GD2.CAR.IL-15 T cells administered to pediatric subjects with relapsed or refractory neuroblastoma or relapsed/refractory osteosarcoma | 4 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (AEs) (CTCAE, version 5.0), a descriptive terminology which can be utilized for AE reporting. A grading (severity) scale is provided for each AE term/symptom: Grade 1 (Mild; asymptomatic); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization indicated; disabling); Grade 4 (Life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to AE). Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).

SECONDARY OUTCOMES:
Identify the maximum tolerated dose (MTD) of iC9.GD2.CAR.IL-15 T cells administered to pediatric subjects with relapsed or refractory neuroblastoma or relapsed/refractory osteosarcoma | 4 weeks
  Tolerability of iC9.GD2.CAR.IL-15 T cells will be assessed by NCI-CTCAE criteria and the CRS grading criteria outlined in Section 12.4 and neurotoxicity/ICANS will be graded according to criteria outlined in Section 12.5
Expansion and persistence of iC9.GD2.CAR.IL-15 cells in vivo | 15 years
  Persistence of iC9.GD2.CAR.IL-15 T cells in vivo will be determined by quantitative Polymerase chain reaction (PCR) and flow cytometry in peripheral blood samples
Anti-tumor response rate to iC9.GD2.CAR.IL-15 t cell administration in pediatric subjects with relapsed or refractory neuroblastoma per Revised International Neuroblastoma Response Criteria (INCR) or relapsed/refractory osteosarcoma by RECIST v1.1 | 6 weeks
  The overall response rate (ORR = complete (CR) + partial (PR) + minor (MR) responses) to iC9.GD2.CAR.IL-15 T cell infusion will be determined using the revised International Neuroblastoma Response Criteria (INRC) for subjects with neuroblastoma. The overall response rate (ORR = complete (CR) + partial (PR) responses) for subjects with osteosarcoma will be measured using Response evaluation criteria in solid tumors (RECIST) version 1.1
Overall survival (OS) in pediatric subjects with relapsed or refractory neuroblastoma or relapsed/refractory osteosarcoma treated with iC9.GD2.CAR.IL-15 T cells | 15 years
  OS will be measured from the date of administration of iC9.GD2.CAR.IL-15 T cells to the date of death
Progression free survival (PFS) in pediatric subjects with relapsed or refractory neuroblastoma or relapsed/refractory osteosarcoma treated with iC9.GD2.CAR.IL-15 T cells | 15 years
  PFS is defined from the date of administration of iC9.GD2.CAR.IL-15 T cells to the date of signs and symptoms of treatment failure or relapse from CR or PR, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: George Hucks, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Emory - Winship Cancer Institute, Atlanta, Georgia
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/patientcare/clinical-trials/